CLINICAL TRIAL: NCT00481429
Title: Evaluation of Predictive Markers of Glitazone Efficacy in Diabetic Patients - Pilot Study
Brief Title: Predictive Markers of Glitazone Efficacy in Diabetic Patients - Pilot Study
Status: Withdrawn | Type: Observational
Why Stopped: Unable to recruit enough participants
Sponsor: Imperial College London (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: cro700
Record Dates: First submitted 2007-05-31; First posted 2007-06-01 (Estimated); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Biomarker; Glitazone; Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Rosiglitazone

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma and urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Rosiglitazone
  Interventions: Drug: Rosiglitazone
- 2: Diet control +/- metformin

INTERVENTIONS:
Drug: Rosiglitazone — Rosiglitazone 4mg od, increased to 4mg bg at 4 weeks if HbA1C above 7%.
  Groups: 1

SUMMARY:
Hypothesis:

A cluster of biochemical measurements (biomarkers) predict which diabetic patients will respond to treatment with a therapeutic dose of rosiglitazone over a 12 week treatment period.

Brief Summary:

The purpose of this study is to assess the predictive value of the biomarkers in diabetic patients treated with a full dose of a thiazolidinedione (eg 4mg bid rosiglitazone) for 12 weeks.

Specifically - the questions asked are:

1. Do baseline measurements of a selected panel of biomarkers predict the patients' response to rosiglitazone over 12 weeks?
2. How does the panel of biomarkers change over that 12 week treatment period?

DETAILED DESCRIPTION:
Rosiglitazone (Avandia) is a medicine used to treat type 2 diabetes. It works by increasing the sensitivity of body tissues to insulin.

This pilot study will examine the possibility that baseline biochemistry might predict the response to rosiglitazone. The study will be conducted in males and the biomarkers of interest measured by specific assays. In addition, since the biomarkers to be measured come from body fat, interpretation of the data would be facilitated by accurate measurements of changes in body fat mass during treatment and these data can be obtained from Echo-MRI scans.

ELIGIBILITY:
Inclusion Criteria:

1. Male subjects aged 18 to 65 years.
2. Eligible subjects must be free from clinically significant illness or disease (other than type 2 diabetes)with the exception of chronic stable-treated hypertension (BP<160/90, and >90/50), thyroid disease (TSH in the normal reference range) and/or dyslipidaemia.
3. BMI must be > or = 25kg/m2 to < or = 40kg/m2,
4. HbA1c between 7and 10%, fasting blood glucose above 7mmol/L (fasting means greater or = 8 hours prior to screening).
5. On diet alone or diet plus metformin (GSK data indicate that the latter group more faithfully reflect the behaviour of 'naive' patients than those who have been washed off prior medications)for at least 1 month.
6. On stable doses of anti-hypertensive medication, thyroid hormone replacement and statin therapy as required.

Exclusion Criteria:

1. Prior treatment with thiazolidinedione, insulin or GLP-1 analogue (Byetta)
2. History of hepatic disease, impairment or abnormal liver function test i.e. AST, ALT>2 times upper limit of normal range (ULN), bilirubin>1.5 time ULN.

   History of renal disease or serum creatinine greater than 1.5 X ULN.
3. Contraindications to rosiglitazone treatment.
4. Serum creatinine greater than 1.5 X upper limit of normal range.
5. Any other clinically significant laboratory abnormality.
6. Claustrophobic or other contraindication to MRI scan
7. Females of child-bearing age who are unwilling to use appropriate methods of contraception.
8. Unable to give informed consent.
9. Unable to comply with study protocol.
10. Clinically significant co-morbidity. -

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with type 2 diabetes attending clinic
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2007-05 (Estimated); Primary Completion 2008-01 (Estimated); Study Completion 2008-01 (Estimated)

PRIMARY OUTCOMES:
The performance of baseline biochemical biomarkers in plasma and urine in distinguishing patients who respond to rosiglitazone from those that do not, as classified by a change in HbA1C at 12 weeks. | 12 weeks

SECONDARY OUTCOMES:
Variability in baseline levels of key biochemical markers in diabetic patients. | 12 weeks
Effect of treatment on a variety of other novel potential predictive biomarkers and markers of insulin sensitisation in diabetic patients. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Martin R Wilkins, MD FRCP, Principal Investigator — Imperial College London
Locations (4):
- United Kingdom (4):
  - Addenbrooke's Hospital, Cambridge
  - Ealing Hospital, London
  - Imperial College London - Hammersmith Campus, London
  - Charing Cross Hospital, London

IPD SHARING:
Plan to Share IPD: No